CLINICAL TRIAL: NCT02815345
Title: Determination by a Noninvasive Method of the Geometric Dimensions of the Nasal Cavities of the Premature Newborn
Brief Title: Objectives and Measures Dimensions Nasal Resistance of Preterm and Term (MODERN)
Acronym: MODERN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Claude Danan, Doctor, Centre Hospitalier Intercommunal Creteil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHIC MODERN
Record Dates: First submitted 2016-05-03; First posted 2016-06-28 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Nose Deformities, Acquired
MeSH Terms: conditions — Nose Deformities, Acquired | interventions — Rhinometry, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measure of the nasal cavity (Experimental): The nasal cavity of all the included neonates will be measured using rhinometry during their hospitalization every weeks. So one to 8 measurement will be performed for each neonates.
  Some included neonates will also have rhinomanometry measurements.
  Interventions: Device: Rhinometry

INTERVENTIONS:
Device: Rhinometry — An acoustic rhinometry device will be used to evaluate the area and the volume of the nasal cavities. Both nasal cavities will be measured except for patients with nasogastric tube.

SUMMARY:
During the resuscitation of preterm infants, withdrawal of non-invasive ventilation is difficult. In a recent study in children gestational age <30 weeks of amenorrhea (SA), definitive withdrawal rate from the first attempt to stop the non-invasive ventilation was 32% . In the same study, the median number of attempts before achieving a final withdrawal was 3 for children born before 28 weeks. The reasons for weaning failure are multiple and little studied. It seems that the type of interface used, mask or cannula, having an influence on the effectiveness of non-invasive ventilation . The nasal lesions induced by non-invasive ventilation are not uncommon, regardless of the interface used . In a recent randomized trial, they ranged from 40% to 50% depending on the type of nasal cannula and non-invasive ventilation mode. It is in this case external damage. But we assume that the breakdown causes internal lesions dependent on the pressure, humidity and flow. These factors are likely to generate a nasal obstruction, source intervention nurses who aspire nasal passages more or less traumatic.

The nasal cavities are often abused and, because of their key role in breathing, could be involved in the withdrawal of ventilatory failure

DETAILED DESCRIPTION:
The measurements of the nasal cavity dimensions are carried out by acoustic rhinometry (about 10 seconds for an acquisition). Measurement of nasal resistance is performed by rhinomanometry earlier (about a minute to a measure). They may be made to wakefulness or sleep since they do not require their participation. These measures will be carried at birth and then every 7 to 10 days (before the age of 28 days), if the child is still hospitalized.

During these measurements, the heart rate and oxygen saturation are collected by a measuring sensor transcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to social security

  * Informed Parental Consent
  * Newborns term and preterm
  * Age less than or equal to 28 days
  * Signature of informed consent by both parents

Exclusion Criteria:

* craniofacial malformation

  * Dyspnea (Silverman score> 3)
  * severe sepsis
  * life-threatened

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Minimal cross sectional area measured by acoustic rhinometry | during the hospitalization of the infants, from birth to week 8
  Acoustic rhinometry is a functional non-invasive procedure based on the sound reflection of acoustic waves on the nasal cavities. This procedure allows determining the geometry and the size of nasal cavities. The device is composed by a wave tube connected to a sound generator emitting series of acoustic impulsions. On this wave tube are laterally connected 2 microphones, themselves connected with a computer which analyzes the acoustic signal. These microphones detect the acoustic reflected wave.

CONTACTS AND LOCATIONS:
Overall Officials: Claude CD DANAN, MD, Principal Investigator — CHI Créteil Neonatalogy
Locations (1):
- CHI CRETEIL Neonatalogy, Créteil, France

IPD SHARING:
Plan to Share IPD: No